CLINICAL TRIAL: NCT07156682
Title: A Single-Arm, Exploratory Study of Iparomlimab and Tuvonralimab (QL1706) Plus XELOX as Neoadjuvant Therapy in Patients With Microsatellite Stable (pMMR/MSS) Resectable Stage III Colon Cancer
Brief Title: QL1706 Plus XELOX as Neoadjuvant Therapy for MSS/pMMR Clinical Stage III Colon Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jing Hao, Deputy Director, Department of Oncology, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202502-005-1
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; MSS/pMMR; QL1706
Keywords: Iparomlimab and Tuvonralimab; QL1706; Neoadjuvant; MSS/pMMR; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 + XELOX (Experimental)
  Interventions: Drug: QL1706; Drug: XELOX

INTERVENTIONS:
Drug: QL1706 — neoadjuvant administered at a dose of 5 mg/kg, intravenous infusion, every three weeks (Q3W), on day 1 of each cycle, 4 cycles
Drug: XELOX — Oxaliplatin 130 mg/m² by intravenous infusion on Day 1; Capecitabine 850-1000 mg/m² orally twice daily (morning and evening) from Day 1 to Day 14; 4 Cycles in total.

SUMMARY:
This is a single-arm, exploratory study enrolling participants with resectable stage III pMMR/MSS colon cancer. Eligible participants who provide written informed consent will receive four cycles of neoadjuvant treatment with iparomlimab and tuvonralimab (QL1706) plus XELOX regimen administered every three weeks (Q3W), followed by radical surgery within two weeks after the last neoadjuvant treatment. After surgery, participants will enter the follow-up phase, or clinicians may decide to administer four additional cycles of adjuvant XELOX chemotherapy based on postoperative pathological findings. The primary endpoint of this study is the pathological complete response (pCR) rate as assessed by investigators. Other endpoints include pathological response (PR), major pathological response (MPR), clinical complete response (cCR), event-free survival (EFS), overall survival (OS), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Histologically or clinically confirmed initially resectable Stage III colon cancer according to the AJCC 8th edition.
* ECOG performance status of 0 or 1.
* pMMR/MSS status confirmed by a local testing center.
* No planned neoadjuvant radiotherapy.
* Participants must voluntarily participate in the study, sign an informed consent form, and demonstrate good compliance.
* Adequate organ function.

Exclusion Criteria:

* Stage IV colon cancer.
* Prior treatment with immune checkpoint inhibitors targeting CTLA-4, PD-1, or PD-L1.
* Current participation in another clinical trial and receiving investigational drugs.
* History of or contraindication to severe allergic reactions to immunotherapy.
* Pregnancy or lactation.
* Active infection requiring treatment.
* Use of immunosuppressive medications.
* Active cardiovascular disease, including stroke or myocardial infarction within 6 months before enrollment, unstable angina, congestive heart failure, or severe uncontrolled arrhythmia requiring medication that may preclude surgery.
* Patients with acute conditions such as obstruction, hemorrhage, or perforation that require immediate surgery.
* Any other condition deemed by the investigator to render the participant unsuitable for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Approximately 1 month after surgery.
  No residual viable tumor cells were found in the postoperative pathological assessment.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | Approximately 1 month after surgery.
  Postoperative pathology shows at least 10% tumor regression.
Pathological Response (PR) | Approximately 1 month after surgery.
  Postoperative pathology shows at least 50% tumor regression.
Clinical Complete Response (cCR) | Approximately 4 months after last participant enrollment.
  No evidence of residual tumor is found via imaging, endoscopic examination, and clinical assessment
Event-Free Survival (EFS) | Approximately 2 years after last participant enrollment.
  The time from initial treatment to the occurrence of any event, including disease progression, treatment discontinuation for any reason, or death.
Overall Survival (OS) | Approximately 2 years after last participant enrollment.
  The time from initial treatment to death from any cause
Adverse Event (AE) | Approximately 2 month after surgery.
  Type, incidence, grading (based on NCI-CTCAE v5.0 criteria), and duration of adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Hao, Deputy Director, Department of Oncology, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China